CLINICAL TRIAL: NCT07256353
Title: Clinical Study on the Safety and Efficacy of Allogeneic, Umbilical Cord Blood Derived CAR T-cell Therapy for B Cell Acute Lymphoblastic Leukemia
Brief Title: Allogeneic UCB-derived CAR-T for B-ALL
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The General Hospital of Western Theater Command (Other)
Collaborators: Chengdu Ucello Biotechnology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yihai2024, Head of Hematology, The General Hospital of Western Theater Command
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YI_UCAR-T_B-ALL_01
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: B-Cell Acute Lymphoblastic Leukemia, Adult
Keywords: allogeneic CAR-T; umbilical cord blood-derived; B-ALL
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UCAR-T cells treatment (Experimental)
  Interventions: Drug: allogeneic umbilical cord blood-derived CAR-T

INTERVENTIONS:
Drug: allogeneic umbilical cord blood-derived CAR-T — intravenous injection of allogeneic umbilical cord blood-derived CAR-T
  Other Names: UCAR-T

SUMMARY:
The purpose of this clinical trial is to learn if allogeneic, umbilical cord blood-derived chimeric antigen receptor T-cell (UCAR-T) therapy works to treat B-cell acute lymphoblastic leukemia (B-ALL) in adults. It will also learn about the safety and efficacy of the allogeneic, umbilical cord blood-derived CAR-T cell product.

The main questions it aims to answer are:

1. What adverse events occur and the incidence rate of dose-limiting toxicities (DLTs) within 28 days and UCAR-T-related adverse events (AEs) after the UCAR-T cell infusion?
2. Which dose level is the optimal biological dose (OBD)?
3. What is the rate of minimal residual disease (MRD) negativity, complete remission (CR) or complete remission with incomplete hematologic recovery (CRi), duration of response (DOR), and overall survival (OS)?

Participants will:

1. May receive lymphodepletion chemotherapy if clinically indicated: fludarabine (30 mg/m²/d, days -5, -4, and -3) and cyclophosphamide (300-500 mg/m²/d, days -5 and -4).
2. If lymphodepletion chemotherapy is administered, rest for 2 days on Day -2 and Day -1.
3. Receive UCAR-T cells infusion on Day 0.
4. Be hospitalized for at least 7 days post-infusion for close safety monitoring and remain within 2 hours of the treatment facility for at least 28 days.
5. Visit the clinic at Day 7, Day 14, Day 28, then monthly for up to 12 months after UCAR-T cells infusion, with continued long-term follow-up for safety and persistence.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years inclusive at the time of signing informed consent.
* Documented diagnosis of B-cell acute lymphoblastic leukemia (B-ALL) according to the National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines in Oncology for Acute Lymphoblastic Leukemia (2018, Version 1) or World Health Organization (WHO) classification criteria.
* CD19 expression or CD20 confirmed by flow cytometry, immunohistochemistry, or pathology on bone marrow, peripheral blood, or tissue specimens. For patients for whom current sampling is not clinically feasible, results from testing performed within 60 days prior to informed consent may be acceptable, as determined by the investigator.
* Life expectancy ≥8 weeks in the opinion of the investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status score <4.
* Adequate organ function as demonstrated by the most recent assessment during the screening period, defined as:

  * Creatinine clearance ≥60 mL/min (calculated using the Cockcroft-Gault formula)
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 × upper limit of normal (ULN)
  * Total bilirubin ≤- 1.5 × ULN (for patients with documented Gilbert's syndrome, total bilirubin ≤- 2.5 × ULN is acceptable)
* For women of childbearing potential (WOCBP), a negative serum pregnancy test must be documented within 7 days prior to enrollment. WOCBP and male patients with partners who are WOCBP must agree to use highly effective contraceptive methods from the screening period through 12 months after CAR-T cell infusion. Women are considered not of childbearing potential if they are postmenopausal for at least 1 year or have documented evidence of surgical sterilization or congenital infertility. Women who are pregnant or breastfeeding are excluded from this study.
* Ability to understand and willingness to provide written informed consent prior to initiation of any study-specific procedures.
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures, including long-term follow-up for up to 15 years.

Exclusion Criteria:

* Active central nervous system (CNS) involvement by B-ALL, defined as CNS-2 or CNS-3 status according to standard criteria.
* History of another malignancy within 2 years prior to screening, except for adequately treated basal cell or squamous cell carcinoma of the skin, or carcinoma in situ of the cervix.
* Patients who previously received CAR-T cell therapy and experienced Grade ≥4 cytokine release syndrome (CRS) or neurotoxicity are specifically excluded.
* Treatment with any investigational or approved anti-B-ALL therapeutic agent within 5 half-lives prior to enrollment (excluding supportive care medications).
* Radioimmunotherapy or radiotherapy within 8 weeks prior to enrollment.
* Receipt of live attenuated vaccine within 4 weeks prior to screening.
* Current or anticipated use of systemic corticosteroids at high dose (defined as a total cumulative dose equivalent to ≥60 mg dexamethasone or equivalent corticosteroid) within 4 weeks prior to lymphodepletion chemotherapy. Physiologic replacement doses, topical, inhaled, nasal, and ophthalmic corticosteroids are permitted.
* Active acute or chronic graft-versus-host disease (GVHD) requiring systemic treatment within 4 weeks prior to CAR-T cell infusion.
* Major surgical procedure within 3 months prior to screening.
* Active CNS disorder or history of irreversible severe CNS toxicity from prior B-ALL therapy resulting in organic brain lesions or CNS dysfunction, including but not limited to seizure disorder, cerebrovascular accident, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis.
* History of hypertensive crisis or hypertensive encephalopathy within 3 months prior to screening.
* Any uncontrolled cardiovascular disease within 6 months prior to enrollment, or any of the following:

  * Ventricular or atrial arrhythmia ≥Grade 2
  * Bradycardia ≥Grade 2
  * Myocardial infarction
  * Severe or unstable angina pectoris
  * Symptomatic congestive heart failure
  * Cerebrovascular accident or transient ischemic attack
  * Pulmonary embolism
  * Deep vein thrombosis
  * Poorly controlled hypertension despite standard medical management
  * Left ventricular ejection fraction (LVEF) <45% as assessed by echocardiography or multigated acquisition (MUGA) scan at screening Pulmonary Exclusions
* Any uncontrolled pulmonary disease within 6 months prior to enrollment, or any of the following:

  * Pulmonary embolism
  * Chronic obstructive pulmonary disease
  * History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis
  * Evidence of active pneumonia on chest computed tomography (CT) scan at screening
  * Symptomatic or uncontrolled interstitial lung disease
  * Clinically significant pulmonary function abnormalities Note: History of radiation pneumonitis/pulmonary fibrosis in a radiation field is permitted if asymptomatic.
* Active bacterial, fungal, protozoal, or viral infection that is not adequately controlled despite appropriate therapy at the time of enrollment, or positive blood culture within 7 days prior to enrollment.
* Known active infection with any of the following:

  * Hepatitis B virus (HBV): Positive HBV surface antigen (HBsAg) or HBV core antibody (HBcAb) with detectable HBV DNA above the normal range
  * Hepatitis C virus (HCV): Positive HCV antibody with detectable HCV RNA above the normal range
  * Human immunodeficiency virus (HIV): Positive HIV antibody
  * Human T-lymphotropic virus (HTLV): Positive HTLV antibody
  * Treponema pallidum (syphilis): Positive T. pallidum antibody
  * Cytomegalovirus (CMV): Positive CMV DNA by polymerase chain reaction (PCR)
* Legally incapacitated individuals under guardianship or conservatorship.
* Psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study or ability to provide informed consent.
* Any abnormal finding, medical condition, or laboratory test result during screening that, in the investigator's judgment, may jeopardize patient safety or interfere with study conduct or interpretation of results.
* Any planned medical or surgical intervention that would interfere with the conduct of the study.
* Contraindication to any medication that may be required during the study, including but not limited to lymphodepletion chemotherapy agents (fludarabine, cyclophosphamide) and medications for management of adverse reactions (e.g., tocilizumab for CRS management, corticosteroids for ICANS management).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence rate of Dose limited toxicity (DLTs) | Up to 28 days after infusion
  Dose limited toxicity(DLT) was defined as the occurrence of any of the following adverse events within 28 days of the infusion of UCAR-T cells.
the rate of adverse events | Up to 28 days after injection
  The number, frequency, severity, and laboratory findings of all treatment-related adverse events/serious adverse events are included.

SECONDARY OUTCOMES:
the rate of minimal residual disease (MRD) negativity | up to 1 year after UCAR-T cells infusion
overall response rate (ORR) | up to 1 year after UCAR-T cells infusiion
Duration of Response (DOR) | up to 1 year after UCAR-T cells infusion
overall survival (OS) | up to 1 year after UCAR-T cells infusion

CONTACTS AND LOCATIONS:
Overall Officials: Hai Yi, M.D. & Ph.D., Principal Investigator — The General Hospital of Western Theater Command
Locations (1):
- The General Hospital of Western Theater Command, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
safety and efficacy data will be shared in a publication.